CLINICAL TRIAL: NCT01377987
Title: Physiological Study to Predict Successful Sleep Apnea Treatment With Acetazolamide in Heart Failure Patients
Brief Title: Predicting Successful Sleep Apnea Treatment With Acetazolamide in Heart Failure Patients
Acronym: HF-ACZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Andrew Wellman (Other)
Collaborators: American Heart Association (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, David Andrew Wellman, Associate Professor of Medicine, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011-P-000049/1
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Heart Failures
MeSH Terms: conditions — Heart Failure | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetazolamide (Experimental)
  Interventions: Drug: Acetazolamide
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — 4 mg/kg, once daily before bed, for 7 days
  Other Names: Diamox
  Arms: Acetazolamide
Drug: Placebo — 4 mg/kg, once daily before bed, for 7 days
  Arms: Sugar pill

SUMMARY:
The ultimate goal is to improve our understanding of the pathophysiology and resistance to effective treatment of sleep disordered breathing in patients with heart failure, with a focus on selecting patients that will benefit specifically from acetazolamide treatment.

The study addresses three primary hypotheses: 1) Acetazolamide treatment will reduce the apnea-hypopnea index and improve markers of heart-failure severity in heart-failure patients with sleep apnea. 2) Acetazolamide will provide the greatest improvement in patients with the most severe ventilatory control instability (strongest chemoreflex response to carbon dioxide; highest loop gain). 3) Acetazolamide will act primarily via stabilizing ventilatory control (reducing loop gain), rather than via improvement to upper airway anatomy, pulmonary congestion, and cardiac function.

ELIGIBILITY:
Inclusion Criteria (Heart failure patients)

* Left ventricular ejection fraction (EF) <50%, or heart failure with preserved EF
* Age 18-89

Exclusion Criteria:

* severe obstructive respiratory disease
* unstable heart failure status
* recent use of positive airway pressure therapy
* current use of opioids, benzodiazepines
* severe kidney disease
* severe anemia

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wellman, MD, PhD, Principal Investigator — Brigham and Women's Hospital; Atul Malhotra, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetazolamide First, Then Placebo: Acetazolamide: 4 mg/kg, once daily before bed, for 7 days
  1 week washout Placebo: 4 mg/kg, once daily before bed, for 7 days
- Placebo First, Then Acetazolamide: Placebo: 4 mg/kg, once daily before bed, for 7 days
  1 week washout Acetazolamide: 4 mg/kg, once daily before bed, for 7 days
Period: First Intervention (7 Days)
Arm/Group | Acetazolamide First, Then Placebo | Placebo First, Then Acetazolamide
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | Acetazolamide First, Then Placebo | Placebo First, Then Acetazolamide
Started | 14 | 15
Completed | 13 | 14
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention (7 Days)
Arm/Group | Acetazolamide First, Then Placebo | Placebo First, Then Acetazolamide
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomized
Groups:
- All Patients: All patients randomized
Arm/Group | All Patients
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Severity of Sleep Disordered Breathing (Apnea-hypopnea Index, AHI)
Description: The frequency of apneas and hypopneas (apnea-hypopnea index) was assessed. The primary measure was the value for non-REM supine sleep. A higher value indicates more severe sleep apnea. A value above 15 indicates the presence of moderate-to-severe sleep apnea.
Time Frame: 1 week
Population: All participants who were randomized and completed the relevant study arm. Data are for non-REM supine sleep.
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- Acetazolamide: Acetazolamide (active arm)
- Placebo: Placebo arm
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 28 | 28
events per hour
  All participants | 26.3 (22.7) | 36.1 (27.8)
  Patients with sleep apnea: number analyzed (Participants) | 22 | 22
  Patients with sleep apnea | 32.3 (22.1) | 44.6 (25.3)

2. Secondary Outcome: Ventilatory Chemoreflex Sensitivity, "Loop Gain" Using Carbon Dioxide Pulses
Description: Chemoreflex "loop gain" was assessed according to Sands SA et al AJRCCM 2017 Jan 15;195(2):237-246. Loop gain is a unitless ratio measure that describes the magnitude of the increase in ventilation that occurs in response to a prior reduction in ventilation ("disturbance") and has units of L/min per L/min. A larger value indicates a more sensitive and unstable control system predisposing to oscillatory breathing. Loop gain was measured on the time scale of 1 min (i.e. response to a 1 cycle/min sinusoidal disturbance, referred to as "LG1"). The procedure involved brief administration of 7% carbon dioxide in air for 0.5 min ("pulses"); tests were repeated every 3 min for 30 min while measuring ventilation and carbon dioxide levels at the nose with patients awake and supine.
  measured using 0.5 min pulses of carbon dioxide.
Time Frame: 1 week
Population: All participants who completed the relevant arm. Morning data are reported.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 28 | 28
unitless | 0.40 (0.16) | 0.49 (0.14)

3. Secondary Outcome: Sympathetic Activity (Urinary Norepinephrine)
Description: Urinary norepinephrine levels overnight
Time Frame: 1 week
Population: All participants who completed the relevant study arm
Measure: Mean (Standard Deviation); unit: ug/g-creatinine
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 28 | 28
ug/g-creatinine | 40.8 (23.6) | 35.0 (17.3)

4. Secondary Outcome: Left-atrial Volume
Description: Left-atrial volume index, echocardiography, bi-plane method. Lower values were considered a favorable outcome. We considered values ≤28 mL/m^2 to indicate normal left atrial volume. Values indicating graded left atrial enlargement were described as follows: mild (29-33 mL/m^2), moderate (34-39 mL/m^2), severe (≥40 mL/m^2).
Time Frame: 1 week
Population: echocardiography could not be performed on one study due to rescheduling issues
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 27 | 28
mL/m^2 | 34.3 (12.1) | 40.0 (13.5)

5. Secondary Outcome: Brain Natriuretic Peptide (NT-proBNP)
Description: Brain natriuretic peptide (NT-proBNP) in morning
Time Frame: 1 week
Population: All participants who completed the relevant arm
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 28 | 28
pg/ml | 919 (1320) | 932 (1403)

6. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: Pittsburgh Sleep Quality Index is a measure of self-reported sleep quality containing 19 questions that make up 7 component scores that are added to provide a total score. Total scores range from 0-21 (units on a scale) with higher scores representing reduced sleep quality. A score of 5 or more is interpreted as reduced sleep quality. The total score is reported.
Time Frame: 1 week
Population: All participants who participated in the relevant study arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetazolamide | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale | 6.7 (3.6) | 7.5 (3.8)

ADVERSE EVENTS:
Arm/Group | Acetazolamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 17/28 | 6/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetazolamide (N=28) | Placebo (N=28)
Fall without injury (General disorders) | 1 (1) | 0 (0) — Fall without injury during 7 days using study medication
Nocturia (Renal and urinary disorders) | 12 (12) | 1 (1) — Self-reported incident nocturia during 7 days using study medication
Taste Disturbance (Metabolism and nutrition disorders) | 4 (4) | 0 (0) — Self-reported incident taste disturbances during 7 days using study medication
Paresthesias (Nervous system disorders) | 5 (5) | 0 (0) — Self-reported incident paresthesias during 7 days using study medication
Fatigue (General disorders) | 3 (3) | 1 (1) — Self-reported incident fatigue during 7 days using study medication
Lightheadedness upon standing (Vascular disorders) | 1 (1) | 1 (1) — Self-reported incident lightheadedness upon standing during 7 days using study medication
Headache (General disorders) | 0 (0) | 1 (1) — Self-reported incident headache during 7 days while using study medication
Gastrointestinal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) — Self-reported incident gastrointestinal discomfort during the 7 days while using study medication
Dry eyes (Eye disorders) | 1 (1) | 0 (0) — Self-reported incident dry eyes during 7 days while using study medication
Reduced exercise tolerance (General disorders) | 0 (0) | 1 (1) — Self-reported incident reduction in exercise tolerance during the 7 days while using study medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No